CLINICAL TRIAL: NCT03564288
Title: A Phase 1 Dose Escalation Trial of SKI-G-801 in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: Study to Find a Safe and Effective Dose of SKI-G-801 in the Treatment of Patients With Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oscotec Inc. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSCO-P1301
Record Dates: First submitted 2018-05-03; First posted 2018-06-20 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2022-05

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation Cohort (Experimental): To identify the recommended phase 2 dose (RP2D) of SKI-G-801 in patients with relapsed or refractory AML (Acute Myeloid Leukemia)
  Interventions: Drug: SKI-G-801

INTERVENTIONS:
Drug: SKI-G-801 — SKI-G-801 is administered as an IV infusion over 10 minutes

SUMMARY:
This Phase I study is designed to assess the safety, tolerability, pharmacokinetics and anti-tumor effect of increasing doses of study drug SKI-G-801 in patients with relapsed or refractory Acute Myeloid Leukemia (AML) who are unresponsive to currently available therapies. Eligible participants will receive cycles of treatment involving IV infusion of SKI-G-801 daily for 14 days followed by 14 days off. Treatment cycles will be repeated until progressive disease or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent for participation, prior to completing any study-related procedures.
* Diagnosis of Acute Myeloid Leukemia (AML)
* Patients must have been off previous antileukemia therapy for at least 2 weeks or 5 half-lives, whichever is longer if the immediate prior regimen included only weekly chemotherapy; or 4 weeks or 5 half-lives, whichever is longer, from any therapy with therapeutic biologics and from any type of investigational therapy. Daily hydroxyurea for up to 2 weeks to keep the absolute blast count below 50 x 10⁹/L will be allowed, but must be discontinued 24 hours prior to administration of study drug. Hydroxyurea will be permitted during the first cycle of treatment if necessary.
* At least one prior induction regimen (with or without consolidation) which may have included hematopoietic stem cell transplantation (HSCT).
* Have adequate liver function.
* Have adequate renal (kidney) function.
* Female patients must either be of non-childbearing potential, or, if of childbearing potential, have a negative urine pregnancy test at screening and agree not to try to become pregnant during the study and for 45 days after the final study drug administration. Women of childbearing potential, if heterosexually active, must agree to use 2 forms of highly effective birth control as determined by the protocol, starting at screening, throughout the study period and for 45 days after the final study drug administration.
* Female patients must agree not to breastfeed at screening, throughout the study period and for 45 days after the final study drug administration.
* Male patients with female spouse/partner of childbearing potential, must agree to use 2 forms of highly effective birth control as determined by the protocol, starting at screening, throughout the study period and for 45 days after the final study drug administration.

Exclusion Criteria:

* Patient has a diagnosis of Acute Promyelocytic Leukemia (APL) or chronic myelogenous leukemia in blast crisis.
* If patient is post allogenic transplant and requires therapy for graft vs host disease (GVHD) within 14 days prior to date of screening.
* Requires treatment with concomitant drugs that prolong QT/QTc interval.
* Recent history of cardiac ischemic disease (acute myocardial infarction within 6 months; uncontrolled angina); severe uncontrolled ventricular arrhythmia; recent transient ischemic attack or stroke within 6 months of screening; poorly controlled hypertension (systolic blood pressure >140 mm Hg or diastolic blood pressure >90 mm Hg).
* Patient has active, untreated central nervous system (CNS) disease.

Other protocol defined inclusion/exclusion criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
Recommended phase 2 dose (RP2D) | From Cycle 1, Day 1 until disease progression, unacceptable toxicity, patient withdrawal from study, or judged not to be in patient's interest to continue in study, assessed up to 36 months
  RP2D of SKI-G-801 determined using Neuenschwander's continual reassessment method (N-CRM)
Patients in complete remission or showing partial response (overall response rate [ORR]) | Up to 30 days following last dose of study drug
  Number of patients showing composite complete remission (complete remission [CR], complete remission with incomplete platelet recovery [CRp], and complete remission with incomplete hematologic recovery [CRi]) of SKI-G-801 according to the Response Criteria in AML
Patients in complete remission | Day 84 (± 3 days)
  Number of patients showing complete remission (CR)
Duration of remission | From date of first reported status of CR to the date of disease relapse or death (+ 1 day); or to date of last available disease status report for patients who do not relapse, assessed up to 36 months
  Number of days between a patient's first reported status of complete remission (CR) and the earlier of disease relapse or death from any cause
Duration of event free survival | Day 1 to date of event (first documented treatment failure, relapse from CR or Cri [CR with incomplete hematologic recovery], or death due to any cause), assessed up to 36 months
  Number of days between start of treatment to date of event
Time to treatment response (TTR) | Day 1 to date of first subsequent disease status of CR (+ 1 day), assessed up to 36 months
  Number of days between the start of treatment to the date of first subsequent disease status of complete remission (CR)
Dose limiting toxicity (DLT) Adverse Events (AEs) | Up to Day 28
  Number of any DLT AEs within the first cycle of each patient's treatment with SKI-G-801

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 30 days following last dose of study drug
  Number, severity (as graded by National Cancer Institute Common Terminology Criteria for Adverse Events [NCI-CTCAE] v4.03), seriousness and relatedness to treatment of treatment-emergent AEs
Number of participants with clinical laboratory abnormalities | Up to 30 days following last dose of study drug
Number of participants with overall safety profiles | Up to 30 days following last dose of study drug
Number of participants with electrocardiogram (ECG) abnormalities | Up to 30 days following last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Eunice Wang, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - USC Norris Comprehensive Cancer Center, Clinical Investigations Support Office (CISO), 1441 Eastlake Ave., Rm. 7327, Los Angeles, California
  - Innovative Clinical Research Institute, Whittier, California

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/